CLINICAL TRIAL: NCT01389076
Title: Phase II Trial of Low-Dose Methotrexate and Iodine I 131 Tositumomab for Previously Untreated, Advanced-Stage, Follicular Lymphoma
Brief Title: Trial of Low-Dose Methotrexate and I 131 Tositumomab for Previously Untreated, Advanced-Stage, Follicular Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Bexxar isn't being produced by the manufacturer as of Feb. 2014
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2010.098; HUM00043235 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Follicular Lymphoma
Keywords: Previously Untreated, Advanced-Stage, Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — tositumomab I-131; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): Low dose methotrexate and Bexxar
  Interventions: Drug: Bexxar; Drug: Low Dose Methotrexate

INTERVENTIONS:
Drug: Bexxar — Iodine I 131 tositumomab (Bexxar) is a radioimmunotherapy (RIT) drug. RIT is a treatment strategy designed to target radiation specifically to cancer cells by attaching a radioactive atom to a monoclonal antibody, an immune system protein that binds to a particular protein. The Iodine I 131 tositumomab (Bexxar) therapeutic regimen is delivered in two sets of intravenous infusions given about 7 days apart. Nonradioactive Tositumomab is given before both the "dosimetric" infusion and the "therapeutic" infusion to improve distribution of these doses throughout the body.
  Other Names: Iodine I 131 tositumomab
Drug: Low Dose Methotrexate — Methotrexate is an antifolate drug. It interferes with cells' ability to copy their DNA. This mainly affects cells that are dividing frequently, such as immune system cells and cancer cells. Methotrexate will be used in this study to try to prevent the occurrence of HAMA by limiting your body's ability to produce anti mouse antibodies.

SUMMARY:
Patients with a type of non-Hodgkin lymphoma, called follicular lymphoma and have not yet had previous systemic treatment, such as chemotherapy or immunotherapy will be invited to participate. This research study is being conducted in order to evaluate the combination of lowdose methotrexate and Iodine I 131 tositumomab (Bexxar) with regards to whether the combination will reduce the occurrence of the HAMA (Human Anti-Mouse Antibody) response. HAMA is an immune reaction against the tositumomab protein. Symptoms arising from HAMA can range from a mild form, like a rash, to a more extreme and possibly life-threatening level. HAMA can also decrease the effectiveness of the treatment, or create a future reaction if a patient is given another treatment containing mouse antibodies. In addition to evaluating the occurrence of HAMA, this research study will also look at the short and long-term effectiveness of this combination in the treatment of lymphoma, as well as its safety.

DETAILED DESCRIPTION:
This is a single-arm, single institution, Phase II study to test the use of low-dose methotrexate in combination with I-131 tositumomab for its ability to lower the rate of (human anti-mouse antibody) HAMA formation in patients with previously untreated low-grade follicular lymphoma. Low-dose methotrexate will be given beginning 3 weeks prior to the first infusion of I-131 tositumomab (4 weekly doses) and continued for 6 weeks (10 total doses), the period of time during which the development of HAMA is most detrimental. A total of 61 patients will be enrolled. The primary endpoint of the study is the determination of the rate of HAMA conversion within the first seven weeks following treatment. The secondary endpoints include response rates, progression-free and overall survival, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically-confirmed diagnosis of follicular non-Hodgkin's B-cell lymphoma, grade 1-2 (grade 1 or grade 2 by WHO classification prior to 2009).
2. Patients must have Ann Arbor Stage III or IV extent of disease after complete staging.
3. Patients must have a willingness and ability to follow prescribed radiation precautions
4. Patients must not have had any previous treatment for low-grade lymphoma including chemotherapy or radiation. They may be newly diagnosed or observed without treatment after diagnosis. Symptomatic and asymptomatic patients will be eligible.
5. Patients must have a performance status of 0-2 on the Eastern Cancer Oncology Group (ECOG) scale and an anticipated survival of at least 3 months.
6. Patients must have an absolute neutrophil count >1500 cells/mm3 and a platelet count >100,000 cells/mm3 within 14 days of study entry. These blood counts must be sustained without support of hematopoietic cytokines or transfusion of blood products.
7. Patients must have adequate renal function (defined as serum creatinine <2.0) and hepatic function (defined as total bilirubin <1.5 x ULN and Aspartate Aminotransferase (AST) <3 x ULN) within 14 days of study entry.
8. Patients must have bi-dimensionally measurable disease.

Exclusion Criteria:

1. Patients with follicular Grade 3a or 3b by WHO Classification.
2. Patients with evidence of active infection requiring IV antibiotics at the time of study entry.
3. Patients with New York Heart Association Class III or IV heart disease or other serious illness that would preclude evaluation.
4. Patients with active obstructive hydronephrosis.
5. Patients with prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years.
6. Patients with known HIV infection.
7. Patients with known brain or leptomeningeal metastases.
8. Patients who are pregnant or nursing. Patients of childbearing potential must undergo a pregnancy test within 7 days of study entry and methotrexate is not to be administered until a negative result is obtained. Males and females must agree to use effective contraception for 6 months following the radioimmunotherapy.
9. Patients with previous allergic reactions to iodine. This does not include reacting to IV iodine-containing contrast materials.
10. Patients with previous allergic reactions to methotrexate.
11. Patients who were previously given any monoclonal antibody, regardless of species, for any condition.
12. Detectable serum levels of HAMA.
13. Patients who are concurrently receiving either approved or non-approved (through another protocol) anti-cancer drugs or biologics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kaminski, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Methotrexate and Bexxar: Low dose methotrexate and Bexxar (tositumomab)
  Patients will begin taking methotrexate 7.5 mg orally once weekly 3 weeks prior to initiating I-131 tositumomab, with additional weekly doses once I-131 tositumomab therapy has begun for a total of 10 doses.
  On Study Day 0, patients will receive the IV administration of 450 mg unlabeled tositumomab followed by the IV administration of the dosimetric dose (5 mCi of Iodine I 131 tositumomab).
Period: Overall Study
Arm/Group | Methotrexate and Bexxar
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Methotrexate and Bexxar
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 56 [36 to 74]
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Rate of Early Onset HAMA (Human Anti-mouse Antibody) Conversion Following Treatment
Description: The percentage of patients that experience early onset HAMA conversion following treatment. Early-onset HAMA is defined as antimouse antibody levels (in blood serum) of at least 5 times the level of detection, occurring at or prior to the 7th week of I-131 tositumomab therapy.
Time Frame: 7 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate and Bexxar
Number analyzed (Participants) | 22
percentage of participants | 18.2 [5.2 to 40.3]

2. Secondary Outcome: Percentage of Participants That Respond to Treatment
Description: The overall response rate (PR [partial response] + CR [complete response]) was determined.
  Partial response is defined as the regression of measurable disease with no new sites of disease.
  Complete response is defined as the disappearance of all evidence of disease.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate and Bexxar
Number analyzed (Participants) | 22
percentage of participants | 90.9 [70.8 to 98.9]

3. Secondary Outcome: The Percentage of Participants Alive at 2 Years
Description: Overall survival was examined at 2 years
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate and Bexxar
Number analyzed (Participants) | 22
percentage of participants | 100

4. Secondary Outcome: Median Progression Free Survival (PFS) Time
Description: The median time patients survived without progression.
Time Frame: 2 Years
Population: Due to the withdrawal of Bexxar by the manufacture and failure to find another supplier, the trial was abandoned and follow-up scans were not obtained. Therefore only survival is known. Progression information is not available.
Arm/Group | Methotrexate and Bexxar
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants That Experienced SAEs During Treatment.
Time Frame: Up to week 13
Measure: Number; unit: participants
Arm/Group | Methotrexate and Bexxar
Number analyzed (Participants) | 22
participants | 2

ADVERSE EVENTS:
Arm/Group | Methotrexate and Bexxar
Serious Adverse Events (participants affected / at risk) | 4/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate and Bexxar (N=22)
back pain (Musculoskeletal and connective tissue disorders) | 1
bilateral Arm Pain (Musculoskeletal and connective tissue disorders) | 1
pain (General disorders) | 1
pain due to disease progression (General disorders) | 1
rectal fissures (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate and Bexxar (N=22)
abdominal pain (Gastrointestinal disorders) | 5
achiness - whole body (General disorders) | 1
acne (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
Arterosclerosis calcifications on spine (Musculoskeletal and connective tissue disorders) | 1
back pain (Musculoskeletal and connective tissue disorders) | 2
bad smell (Nervous system disorders) | 1
Bilateral Arm Paresthesias (Nervous system disorders) | 1
Bilateral Foot Swelling (Vascular disorders) | 1
Bilateral Leg Pain (Musculoskeletal and connective tissue disorders) | 1
bleeding gums (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Blood in stool (Gastrointestinal disorders) | 1
bruising (Vascular disorders) | 3
Burning sensation of skin (Nervous system disorders) | 1
Chest Tenderness (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 3
Cholelithiasis (Gastrointestinal disorders) | 1
conjunctivitis (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Decreased ANC (Blood and lymphatic system disorders) | 6
Decreased WBC (Blood and lymphatic system disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Dizziness (Nervous system disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
dysgeusia (Gastrointestinal disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Elevated Creatinine (Investigations) | 1
Facial Flushing (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 8
Fever (General disorders) | 2
Finger Puncture wound (Injury, poisoning and procedural complications) | 1
flu-like symptoms (General disorders) | 1
forgetful (Psychiatric disorders) | 1
General Arthalgias (Musculoskeletal and connective tissue disorders) | 1
General Myalgias (Musculoskeletal and connective tissue disorders) | 1
Generalized Itching (Skin and subcutaneous tissue disorders) | 1
Generalized rash (Skin and subcutaneous tissue disorders) | 1
Hand Paresthesia (Nervous system disorders) | 1
Hand tremor (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypothyroidism (Investigations) | 2
infusion related reaction (Immune system disorders) | 1
Insomnia (Psychiatric disorders) | 1
irritable (Psychiatric disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 3
Jaw pain (Musculoskeletal and connective tissue disorders) | 1
Left hip pain (Musculoskeletal and connective tissue disorders) | 1
Leg pain - bilateral (Musculoskeletal and connective tissue disorders) | 1
loose stool (Gastrointestinal disorders) | 1
Lower extremity neuropathy (Nervous system disorders) | 1
Lower extremity swelling (Vascular disorders) | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1
Mild Narrowing of C3-4, C4-5 (Musculoskeletal and connective tissue disorders) | 1
Muscle Soreness (Musculoskeletal and connective tissue disorders) | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 11
Night sweats (General disorders) | 1
Non-productive cough (Respiratory, thoracic and mediastinal disorders) | 2
numbness hands (Nervous system disorders) | 1
occasional Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Pain around tumor site (General disorders) | 1
Pain in bilateral axilla (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in lower extremities and bilateral groin (Musculoskeletal and connective tissue disorders) | 1
Pain on bilateral feet (Musculoskeletal and connective tissue disorders) | 1
Papular rash on anterior chest (Skin and subcutaneous tissue disorders) | 1
Papular rash on lower neck (Skin and subcutaneous tissue disorders) | 1
Periorbital edema (Eye disorders) | 1
Phonophobia (Psychiatric disorders) | 1
Photophobia (Eye disorders) | 1
Pityriasis Rosea (Skin and subcutaneous tissue disorders) | 1
pleuritic chest pain (Musculoskeletal and connective tissue disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary nodules (Respiratory, thoracic and mediastinal disorders) | 1
Puritus (Skin and subcutaneous tissue disorders) | 1
Rash on tumor site (Skin and subcutaneous tissue disorders) | 1
rash, neck (Skin and subcutaneous tissue disorders) | 1
Rectal bleeding (Gastrointestinal disorders) | 1
Rhinnorhea (Respiratory, thoracic and mediastinal disorders) | 1
Right ankle fracture (Injury, poisoning and procedural complications) | 1
Right leg Pain (Musculoskeletal and connective tissue disorders) | 1
Right Leg Paresthesia (Nervous system disorders) | 1
Right maxillary sinus pain (Respiratory, thoracic and mediastinal disorders) | 1
Scaly rash on upper extremities, bilateral (Skin and subcutaneous tissue disorders) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Sinus infection (Infections and infestations) | 2
sinus pressure (Respiratory, thoracic and mediastinal disorders) | 1
Small scattered ecchymosis on lower extremities (Vascular disorders) | 1
Sore Throat (Gastrointestinal disorders) | 3
Swelling around eyes (Eye disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 6
upper respiratory infection (Infections and infestations) | 3
Urinary Frequency (Renal and urinary disorders) | 1
UTI (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
warm/burning sensation in throat (Nervous system disorders) | 1
wooziness (Nervous system disorders) | 1
Worsening GERD (Gastrointestinal disorders) | 1
yeast infection (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
This trial was abandoned prematurely due to the withdrawal of Bexxar by the manufacturer and failure to find another supplier.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes